CLINICAL TRIAL: NCT06114953
Title: Comparative Efficacy of Mizoribine With Mycophenolate Mofetil for Living Related Kidney Transplantation Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRDN-LEES-2023-10
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Kidney Transplant Immunosuppression
Keywords: Immunosuppression; Kidney Transplant Rejection; mizoribine
MeSH Terms: interventions — mizoribine; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Experimental group: glucocorticoid, mizoribine, tacrolimus; Control group: glucocorticoid, mycophenolate mofetil.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mizoribine group (Experimental): Mizoribine, glucocorticoid, tacrolimus
  Interventions: Drug: Mizoribine
- Mycophenolate group (Active Comparator): Mycophenolate mofetil, glucocorticoid, tacrolimus
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mizoribine — Mizoribine+glucocorticoid+tacrolimus after kidney transplantation
  Arms: Mizoribine group
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil+glucocorticoid+tacrolimus after kidney transplantation
  Other Names: Mycophenolate Acid
  Arms: Mycophenolate group

SUMMARY:
This prospective, randomized controlled study is intended to enroll 152 patients in the early stages of donor kidney transplantation at six clinical centers in China between January 2023 and January 2024. All patients meeting the inclusion criteria were randomly assigned 1:1 to either Mizoribine or Mycophenolate Mofetil for 12 months. At the baseline of follow-up (before enrollment) and each follow-up point, all clinical indicators of patients were recorded to measure the therapeutic effect.

DETAILED DESCRIPTION:
This is a multi-center, prospective, non-inferior, randomized controlled clinical study. The sick individuals and their families participating in the trial voluntarily participate and sign the "informed consent" under the premise of fully understanding the treatment plan; The treatment plan was approved by the hospital ethics committee.

A total of 152 patients from six centers nationwide will be enrolled starting from the date when the center's ethics are officially approved. The qualified recipients of donor kidney transplantation were randomly assigned 1:1 to the control group and the experimental group. The control group was treated with glucocorticoid + MPA+ tacrolimus for 12 months, and the experimental group was treated with glucocorticoid +MZR+ tacrolimus for 12 months. All subjects were followed up on the day of renal transplantation, at 1, 2 weeks and 1, 2, 3, 6, 9 and 12 months after the operation: history collection, incidence of acute rejection, survival rate of recipients, survival rate of transplanted kidney, liver and kidney function, blood routine and urine routine; Cytomegalovirus (CMV)-DNA and BK virus (BKV)-DNA copy levels were detected in blood at 1, 3, 6, 9, and 12 months after renal transplantation to assess CMV and BKV infection. Adverse reactions were recorded during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1) After donor kidney transplantation;
* 2) Adult recipients aged 18-75 years, regardless of gender;
* 3) First-time kidney transplant recipients;
* 4) Voluntarily sign written informed consent.

Exclusion Criteria:

* 1) Multiple organ transplantation;
* 2) DSA positive patients had ABO incompatibility and PRA>30%;
* 3) Recipients with active signs of infection;
* 4) Recipients with leukocyte counts below 3,000/mm3;
* 5) Pregnant women, breastfeeding women or women who do not wish to use appropriate contraceptive methods during the study period;
* 6) Patients with severe gastrointestinal diseases and active peptic ulcer disease;
* 7) suffering from any mental illness;
* 8) Patients with severe heart disease and abnormal heart function;
* 9) Subjects who are known to be allergic to the test drug;
* 10) Recipients judged unsuitable for inclusion by other competent physicians.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine | Postoperative 1 week, 2 weeks, 1month, 2，3，6，9，12 months
  Monitoring serum creatinine.

OTHER OUTCOMES:
White blood cell | Postoperative 1 week, 2 weeks, 1month, 2，3，6，9，12 months.
  Detect the count of white blood cell.
Cytomegalovirus DNA copies. | Postoperative 3，6，12 months.
  Detect Cytomegalovirus DNA copies in blood.
BK Virus DNA copies. | Postoperative 3，6，12 months.
  Detect BK virus DNA copies in blood and urine.
Uric Acid | Postoperative 1 week, 2 weeks, 1month, 2，3，6，9，12 months.
  Check uric acid levels.

CONTACTS AND LOCATIONS:
Overall Officials: TAO LIN, Doctor, Study Chair — West China Hospital
Locations (6):
- China (6):
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - West China Hospital, Sichuan University, Chengdu

IPD SHARING:
Plan to Share IPD: No
No IPD shared plan.

REFERENCES:
- [Result] Shi Y, Liu H, Chen XG, Shen ZY. Efficacy and Safety of Mizoribine Combined With Tacrolimus in Living Donor Kidney Transplant Recipients: 3-Year Results by a Chinese Single Center Study. Transplant Proc. 2019 Jun;51(5):1337-1342. doi: 10.1016/j.transproceed.2019.03.014. PMID 31155174
- [Result] Ju MK, Huh KH, Park KT, Kim SJ, Cho BH, Kim CD, So BJ, Kang CM, Lee S, Joo DJ, Kim YS. Mizoribine versus mycophenolate mofetil in combination therapy with tacrolimus for de novo kidney transplantation: evaluation of efficacy and safety. Transplant Proc. 2013 May;45(4):1481-6. doi: 10.1016/j.transproceed.2012.12.028. PMID 23726602
- [Result] Huh KH, Lee JG, Ha J, Oh CK, Ju MK, Kim CD, Cho HR, Jung CW, Lim BJ, Kim YS; RECORD Study. De novo low-dose sirolimus versus mycophenolate mofetil in combination with extended-release tacrolimus in kidney transplant recipients: a multicentre, open-label, randomized, controlled, non-inferiority trial. Nephrol Dial Transplant. 2017 Aug 1;32(8):1415-1424. doi: 10.1093/ndt/gfx093. PMID 28810721
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091